CLINICAL TRIAL: NCT04477967
Title: Children's Hospital of Chongqing Medical University
Brief Title: Design and Implementation of the Pediatric Liver Transplantation Biobank
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qiu Li, dean, Children's Hospital of Chongqing Medical University
Other Study IDs: 2018（120）
Record Dates: First submitted 2020-07-08; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Liver Diseases; Liver Transplant; Complications; Pediatric ALL
MeSH Terms: conditions — Liver Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There are no interventions because it is a protocol study

SUMMARY:
The purpose of the pediatric liver transplant biobank is to systematically collect clinical specimens from pediatric end-stage liver disease. It is expected to contribute to the research and development of paediatric end-stage liver disease in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with end-stage liver disease.
2. Liver transplantation in our hospital.
3. informed patient consent.
4. long-term follow-up in our hospital.

Exclusion Criteria:

No fixed contact information, difficult to follow up the patients.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with end-stage liver disease who undergo liver transplantation in our hospital. Obtain their or their parents' informed consent before the project starts.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Biological sample bank | 2 years
  A repository of biological samples from patients who will join the project, will be organised at the biobank center of the Children's Hospital of Chongqing Medical University(CHCMU) under the responsibility of the experienced staff at the Department of Hepatic.
Integrated health data platform | 2 years
  Collect patient clinical test information and establish diagnostic database.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Xiang Z, Wang R, Lu Y, Li Y, Wang H, Xiong Q, Dai X, Guo H, Deng Y, Le Y, Zhang M, Zhao Y. Study Protocol: Design and Implementation of the Pediatric Liver Transplantation Biobank. Biopreserv Biobank. 2021 Apr;19(2):111-118. doi: 10.1089/bio.2020.0128. Epub 2021 Apr 12. PMID 33847526